CLINICAL TRIAL: NCT01660360
Title: A Phase I Study of the Safety and Pharmacokinetics of a Fully Human Monoclonal Antibody to the Vascular Endothelial Growth Factor Receptor2 (Tanibirumab) in Patients With Advanced Cancers or Metastatic Cancer
Brief Title: Phase I Trial of Tanibirumab in Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmAbcine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMC1101-TAAC01
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: Tanibirumab Phase I trial
MeSH Terms: conditions — Neoplasm Metastasis | interventions — olinvacimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tanibirumab (Experimental): The total dose of Tanibirumab for each patient will depend on dose level assignment and the patient's weight. Dose levels to be potentially tested in Phase I include: 1 mg/kg, 2 mg/kg, 4 mg/kg, 8 mg/kg, 12 mg/kg, 16 mg/kg, and 20 mg/kg.
  Interventions: Biological: Tanibirumab

INTERVENTIONS:
Biological: Tanibirumab

SUMMARY:
The primary objective of this study is to assess the safety, tolerability, and maximum tolerated dose (MTD) of Tanibirumab in patients with advanced or metastatic cancer who are refractory or for whom there are no standard therapeutic option.

* To evaluate the pharmacokinetics of Tanibirumab in such patients
* To determine a recommended phase II dose (RP2D) of Tanibirumab based on above assessments

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, open-label, non-randomized, dose-escalating study of Tanibirumab which is a fully human monoclonal antibody to vascular endothelial growth factor receptor 2 (VEGFR2/KDR). This study will enroll patients with advanced or metastatic cancer who are refractory or for whom there are no standard therapeutic options. Tanibirumab will be administered intravenously to such patients over 60 minutes on Day 1, 8, and 15 (subject to change pending PK and toxicity data). Each treatment cycle will be a minimum of 28 days in length. The dose escalation study employing a 3 + 3 design is designed to identify the RP2D which will be based on safety, tolerability and PK of the RP2D. This study is expected to enroll a total of approximately 18-24 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* Signed informed consent
* Histologically documented, incurable, locally advanced or metastatic cancers that have failed to respond to at least one prior regimen or for which there is no standard therapy.
* Disease that is measurable or evaluable by RECIST 1.1 criteria (for Solid Tumors)
* ECOG performance status 0-2
* Documented negative pregnancy test for women of childbearing potential and use of an effective means of contraception for both men and women while enrolled in the study
* Granulocyte count ≥ 1,500/㎣, platelet count ≥ 100,000/㎣, and hemoglobin ≥ 9 g/dL
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN)(≤ 3 x ULN if liver metastatic cancer)
* Alkline phosphatase, AST and ALT ≤ 2.5 x ULN (≤ 5 x ULN if liver metastatic cancer)
* Serum creatinine ≤ 1.5 mg/dL
* INR (international normalized ratio) ≤ 1.3, and aPTT (activated partial thromboplastin time) ≤ 1.5 x ULN
* Subject had to have a projected life expectancy of at least 3 months
* Bazetts correction QTc < 450 msec in ECG at Screening

Exclusion Criteria:

* Less than 4 weeks since last chemotherapy (including biologic unless previous Avastin treatment, experimental, and hormonal therapy), radiation therapy, or major surgical procedure
* All incisions from any procedure must be fully healed and sutures removed prior to infusion on Day 1
* Pleural effusions, ascites, or leptomeningeal disease as the only manifestation of the current malignancy
* Subjects that have hypertension that is remained uncontrolled, despite drug regimen.
* Subjects with grade III or IV hemorrhage/bleeding and who have experienced pulmonary hemorrhage/hemoptysis (exceed size of 2.5 mL of erythrocyte) or who have experienced grade III/IV hemorrhage/bleeding.
* The presence of gastrointestinal perforation
* The presence of tracheoesophageal fistula or grade Ⅳ fistula
* Subjects with grade Ⅳ proteinuria (nephritic syndrome)
* The presence of arterial thromboembolic events
* Subjects who have history of life threatening (grade Ⅳ) pulmonary embolism
* Subjects with a known hypersensitivity to CHO cell product or other recombined human or humanized antibody
* Subjects with mental illness
* Subjects with a known hypersensitivity to any of the ingredients/substrates in investigational product of this study
* Subjects who given any investigational drug within longer period between 30 days and 5 times of half life before participation in this study
* Active infection requiring IV antibiotics
* Active autoimmune disease that is not controlled by drugs
* Clinically important history of liver disease, including viral or other active hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus (HIV) infection
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the subjects at high risk from treatment complications
* Significant traumatic injury within 3 weeks of Day 1
* Inability to comply with study and follow-up procedures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 28days
  The safety and tolerability of Tanibirumab will be assessed using the following measures: frequency and nature of dose-limiting toxicities (DLTs); nature, severity, and relatedness of adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, v4.0; changes in vital signs; and changes in clinical laboratory parameters.

SECONDARY OUTCOMES:
Pharmacokinetics | Cycle 1 : predose, 0.5, 2, 4, 24 and 72 hours after 1st dose, predose and 0.5 hours after 2nd dose, predose, 0.5, 2, 4, 24, 72, 168 and 336 hours after 3rd dose. After cycle 2: predose of 1st dose and 0.5 hour after 3rd dose.
  The following PK parameters will be derived from the serum concentration-time profile of Tanibirumab following administration: serum total exposure (AUC), Cmax, clearance, volume of distribution (central compartment Vc and at steady state Vss), and half-life (t½).
Efficacy | completion of 2 and more cycle
  The following activity outcome measures will be assessed: objective response, defined as a complete or partial response confirmed 4 weeks after initial documentation; duration of objective response; and progression-free survival. Objective response and disease progression will be determined using RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Young Seok Park, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea